CLINICAL TRIAL: NCT03073902
Title: Clinical Research for the Correlation of PD-L1 Expression in Non-small Lung Cancer Tissue and Peripheral Blood T Cell and Serum.
Brief Title: The Correlation of PD-L1 Expression in Non-small Lung Cancer Tissue and Peripheral Blood T Cell and Serum.
Status: Completed | Type: Observational
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy Director,Head of Oncology department, Principal Investigator, Clinical Professor, Xinqiao Hospital of Chongqing
Other Study IDs: XQonc-006
Record Dates: First submitted 2017-02-26; First posted 2017-03-08 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: NSCLC
MeSH Terms: interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observed group: The project is planned to explore the correlation of PD-L1 expression in non-small lung cancer tissue and peripheral blood T cell and serum.The investigators have designed to detected the expression levels of PD-L1 protein in cancer tissue and detected the expression levels of PD-L1 in peripheral blood T cell and serum by using variance analysis of repeated measures design information.
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — Liquid biopsy

SUMMARY:
The detection of tissue PD-L1 immunohistochemistry in Non-small cell lung cancer (NSCLC) has an important role in guiding for the treatment of immune detection point. At the same time,tissue detection is time-consuming and laborious, liquid biopsy can reflect the information of tumor tissue,PD-L1 expression in serum and peripheral blood T cell are expected to be simple, rapid, non-invasive means of detection. The project is planned to explore the correlation of PD-L1 expression in non-small lung cancer tissue and peripheral blood T cell and serum..The investigators have designed to detected the expression levels of PD-L1 protein in cancer tissue and detected the expression levels of PD-L1 in peripheral blood T cell and serum.By using variance analysis of repeated measures design information. Thus exploring the correlation of PD-L1 expression in non-small lung cancer tissue and peripheral blood T cell and serum,guiding clinical practice of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological histology and/or cytology confirmed non-small lung cancer;
2. Voluntarily enrolled to participate in,better compliance, cooperate with experimental observations, and sign informed consent.

Exclusion Criteria:

1. Vital organs (e.g., heart, liver, kidney) have serious dysfunction;
2. Patients with a history of autoimmune disease;
3. Patients with participating in other clinical trials at the same time;
4. Other cases that researchers believe that patients should not participate in the present trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathological histology and/or cytology confirmed non-small lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
The match rate of PD-L1 protein expression in non-small lung cancer tissue and peripheral blood T cell . | up to two years
  consistency
The match rate of PD-L1 protein expression in non-small lung cancer tissue and serum. | up to two years
  consistency

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiao Hospital of Chongqing, Chongqing, China